CLINICAL TRIAL: NCT04277533
Title: Evaluation of Some Blood Biomarkers as Predictors of Neonatal Necrotizing Enterocolitis
Brief Title: Predictors of Neonatal Necrotizing Enterocolitis
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Esraa Ragab Zaki, DR Esraa Ragab Zaki, Ain Shams University
Other Study IDs: necrotizing enterocolitis
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Necrotising Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: NEC preterm neonates with gestational ages are between 28-36 weeks regardless of birth weight. NEC diagnosis and staging will be according to Bell's staging criteria .
  Interventions: Diagnostic Test: Serum γ-Glutamyl transferase (GGT), Total serum bilirubin (TSB), Serum calcium concentration (Ca2+), Peripheral blood neutrophil to lymphocyte ratio (NLR)
- Control group: Stable preterm neonate with matched gestational and postnatal ages without infectious diseases.
  Interventions: Diagnostic Test: Serum γ-Glutamyl transferase (GGT), Total serum bilirubin (TSB), Serum calcium concentration (Ca2+), Peripheral blood neutrophil to lymphocyte ratio (NLR)

INTERVENTIONS:
Diagnostic Test: Serum γ-Glutamyl transferase (GGT), Total serum bilirubin (TSB), Serum calcium concentration (Ca2+), Peripheral blood neutrophil to lymphocyte ratio (NLR) — GGT, Ca2+, NLR and TSB are serum markers which had been studied for early detection and prediction of severity of NEC.

SUMMARY:
To assess the value of peripheral blood neutrophil to lymphocyte ratio (NLR), serum levels of γ-Glutamyl transferase (GGT), total serum bilirubin and serum calcium (Ca2+) concentrations for early diagnosis and prediction of NEC severity and if found significant, scoring will be done according to their levels in different Bell's stages.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is primarily a disease process of the gastrointestinal tract of neonates that results in inflammation and bacterial invasion of the bowel wall.

Despite extensive research, the pathophysiology of NEC remains unclear and therapeutic options are limited.

Clinical manifestations of NEC may be vague, including increased episodes of apnea, desaturations, bradycardia, lethargy and temperature instability.

There may also be GI-specific symptoms such as feeding intolerance, emesis, bloody stools, abdominal distention and tenderness, and abdominal wall discoloration.

Radiographic signs may include ileus, dilated or fixed intestinal loops, air in the intestinal wall or free air in the abdomen.

NEC diagnosis, however, remains challenging because many now see that Bell's staging criteria currently used for diagnosis as being not accurate.

Neutrophil to lymphocyte ratio (NLR) is used as a marker of subclinical inflammation. It is calculated by dividing the number of neutrophils by number of lymphocytes, usually from peripheral blood sample. Increase of neutrophil proportion just reflects the deterioration of the immune system, while decreased lymphocyte ratio reflects the increasing level of physical stress.

Further NLR is closely related to the inhibition of body's immune function. In a word, NLR could indicate the status of body's inflammation response and the level of physical stress timely and accurately.

In a clinical study conducted in 2001, the authors suggested the routine use of NLR as a stress factor in clinical ICU practice, and they claimed that NLR might has a prognostic and a predictive value of many diseases.

Gamma glutamyl transferase (GGT) is an enzyme found in the cell membranes of many tissues. The highest concentration is in the kidney, but the liver is considered the source of normal enzyme activity. GGT is involved in the transfer of amino acids across the cell membrane and also in leukotriene metabolism. It has an intracellular antioxidant effect because it is involved in glutathione metabolism, resulting in the formation of cysteine. GGT is cleared from the plasma by liver uptake.

Bilirubin is a free radical scavenger with anti-inflammatory and antioxidant property. One report described that stage III NEC had lower total serum bilirubin than their mild or disease-free controls during the first 14 days of life. Since serum bilirubin level is a function of the activity of UGT1A1, albumin binding, and the bilirubin load; it will be important to determine if serum bilirubin concentration correlates with NEC development or severity.

A relatively constant serum calcium (Ca2+) concentration is vital for cellular function and under strict control by the neural/humoral factors. It is unclear what causes serum Ca2+ lower in NEC neonates. In a recent report, higher level of serum GGT, a significantly lower serum bilirubin and Ca2+ were found in severe NEC.

ELIGIBILITY:
Inclusion Criteria:

• Patient group: NEC preterm neonates with gestational ages are between 28-36 weeks regardless of birth weight. NEC diagnosis and staging will be according to Bell's staging criteria.

• Control group: Stable preterm neonate with matched gestational and postnatal ages without infectious diseases will be included.

Exclusion Criteria:

* Neonates with congenital infectious diseases, perinatal asphyxia, severe birth defects, congenital digestive tract malformations, inherited metabolic diseases or parental refusal of enrollment.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates with gestational ages are between 28-36 weeks regardless of birth weight.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of some blood biomarkers as predictors of neonatal necrotizing enterocolitis. | Baseline
  The peripheral blood neutrophil to lymphocyte ratio (NLR), serum levels of γ-Glutamyl transferase (GGT), total serum bilirubin and serum calcium (Ca2+) concentrations would been studied for early diagnosis and prediction of NEC severity and if found significant, scoring will be done according to their levels in different Bell's stages.

CONTACTS AND LOCATIONS:
Overall Officials: Nehal El-Raggal, MD, Study Director — faculty of medicine ain shams university; Dina Essam, Study Director — faculty of medicine ain shams university; Azza Hassan, Study Director — faculty of medicine ain shams university; Yasser Wageih, Study Director — faculty of medicine ain shams university
Locations (1):
- Ain Shams university Faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
I can share my information as a researcher.

REFERENCES:
- [Background] Bell MJ, Ternberg JL, Feigin RD, Keating JP, Marshall R, Barton L, Brotherton T. Neonatal necrotizing enterocolitis. Therapeutic decisions based upon clinical staging. Ann Surg. 1978 Jan;187(1):1-7. doi: 10.1097/00000658-197801000-00001. PMID 413500
- [Background] Cabrera-Abreu JC, Green A. Gamma-glutamyltransferase: value of its measurement in paediatrics. Ann Clin Biochem. 2002 Jan;39(Pt 1):22-5. doi: 10.1258/0004563021901685. PMID 11853185
- [Background] de Jager CP, van Wijk PT, Mathoera RB, de Jongh-Leuvenink J, van der Poll T, Wever PC. Lymphocytopenia and neutrophil-lymphocyte count ratio predict bacteremia better than conventional infection markers in an emergency care unit. Crit Care. 2010;14(5):R192. doi: 10.1186/cc9309. Epub 2010 Oct 29. PMID 21034463
- [Background] Fereshtehnejad SM, Poorsattar Bejeh Mir K, Poorsattar Bejeh Mir A, Mohagheghi P. Evaluation of the possible antioxidative role of bilirubin protecting from free radical related illnesses in neonates. Acta Med Iran. 2012;50(3):153-63. PMID 22418983
- [Background] Gordon PV, Swanson JR, Attridge JT, Clark R. Emerging trends in acquired neonatal intestinal disease: is it time to abandon Bell's criteria? J Perinatol. 2007 Nov;27(11):661-71. doi: 10.1038/sj.jp.7211782. Epub 2007 Jul 5. PMID 17611610
- [Background] Han CQ and Wei XY (2017): Novel biomarkers to determine neonates with necrotizing enterocolitis, Biomedical Research; 28 (13): 6002-6006.
- [Background] Levitt DG, Levitt MD. Quantitative assessment of the multiple processes responsible for bilirubin homeostasis in health and disease. Clin Exp Gastroenterol. 2014 Sep 2;7:307-28. doi: 10.2147/CEG.S64283. eCollection 2014. PMID 25214800
- [Background] Li B, Zhang ZL, Yang ZZ, Zhang HZ. (2012): Application value of neutrophil and lymphocyte count ratio in respiratory tract infectious diseases. Zhong Guo Xue Ye Liu Bian Xue Za Zhi; 22: 522-524. In Chinese.
- [Background] Lin PW, Stoll BJ. Necrotising enterocolitis. Lancet. 2006 Oct 7;368(9543):1271-83. doi: 10.1016/S0140-6736(06)69525-1. PMID 17027734
- [Background] Stocker R, Yamamoto Y, McDonagh AF, Glazer AN, Ames BN. Bilirubin is an antioxidant of possible physiological importance. Science. 1987 Feb 27;235(4792):1043-6. doi: 10.1126/science.3029864.
- [Background] Terrin G, Stronati L, Cucchiara S, De Curtis M. Serum Markers of Necrotizing Enterocolitis: A Systematic Review. J Pediatr Gastroenterol Nutr. 2017 Dec;65(6):e120-e132. doi: 10.1097/MPG.0000000000001588. PMID 28379923
- [Background] Thompson AM, Bizzarro MJ. Necrotizing enterocolitis in newborns: pathogenesis, prevention and management. Drugs. 2008;68(9):1227-38. doi: 10.2165/00003495-200868090-00004. PMID 18547133
- [Background] Yajamanyam PK, Rasiah SV, Ewer AK. (2014): Necrotizing enterocolitis: current perspectives, Dove Medical Press Limited, Volume 2014:4 Pages 31-42
- [Background] Yang M, Li L, Su N, Lin J, Wang J. [Dynamic monitoring of the neutrophil/lymphocyte ratio could predict the prognosis of patients with bloodstream infection]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2015 Jun;27(6):471-6. doi: 10.3760/cma.j.issn.2095-4352.2015.06.011. Chinese. PMID 26049186
- [Background] Yang Y, Cao ZL, Zhou XY, Chen XQ, Pan JJ, Cheng R. Does neutrophil/lymphocyte ratio have good diagnostic value in neonatal necrotizing colitis? J Matern Fetal Neonatal Med. 2019 Sep;32(18):3026-3033. doi: 10.1080/14767058.2018.1455182. Epub 2018 Mar 27. PMID 29557695
- [Background] Yokoyama H. [Gamma glutamyl transpeptidase (gammaGTP) in the era of metabolic syndrome]. Nihon Arukoru Yakubutsu Igakkai Zasshi. 2007 Jun;42(3):110-24. Japanese. PMID 17665541
- [Background] Zahorec R. Ratio of neutrophil to lymphocyte counts--rapid and simple parameter of systemic inflammation and stress in critically ill. Bratisl Lek Listy. 2001;102(1):5-14. English, Slovak. PMID 11723675
- [Background] Zimmerman K., Daniel K. (2018): Principals and practice of pediatric infectious diseases textbook, Chapter H. Gastrointestinal Tract Infections and Intoxications, necrotizing enterocolitis; page 394-397